CLINICAL TRIAL: NCT06374589
Title: Closed-Loop O2 Use During High Flow Oxygen Treatment of Critical Care Adult Patients (CLOUDHFOT)- a Randomized Cross-over Study
Brief Title: Closed-Loop O2 Use During High Flow Oxygen Treatment of Critical Care Adult Patients (CLOUDHFOT)
Acronym: CLOUDHFOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202303123
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Hypoxemic Respiratory Failure; Acute Hypercapnic Respiratory Failure; Respiratory Depression; Respiratory Failure
Keywords: Acute respiratory failure (ARF); HFNC; Closed-loop
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Close-loop FiO2 Controller (Experimental): Six hours period where the fraction of inspired oxygen (FiO2) delivered will be automatically titrated based on SpO2 values obtained from the patient.
  Interventions: Device: Closed-loop FiO2 controller
- Conventional (Active Comparator): Six hours period where the fraction of inspired oxygen (FiO2) delivered will be manually titrated by clinician based on SpO2 values obtained from the patient.
  Interventions: Device: Conventional

INTERVENTIONS:
Device: Closed-loop FiO2 controller — Close-loop FiO2 controller software option provides automated adjustment of the ventilator Oxygen setting to maintain the patient's SpO2 in a defined target range. When using the software option, the user defines the SpO2 target range, as well as the SpO2 emergency limits, and the device adjusts the FiO2 setting to keep the patient's SpO2 in the target range.
  Arms: Close-loop FiO2 Controller
Device: Conventional — Six hours period where the fraction of inspired oxygen (FiO2) delivered will be manually titrated by clinician based on SpO2 values obtained from the patient.
  Arms: Conventional

SUMMARY:
High flow nasal oxygen therapy (HFNO) is an established modality in the supportive treatment of patients suffering from acute hypoxemic respiratory failure. The high humidified gas flow supports patient's work of breathing, reduces dead space ventilation, and improves functional residual capacity while using an unobtrusive patient's face interface [Mauri et al, 2017; Möller et al, 2017].

As hyperoxia is considered not desirable [Barbateskovic et al, 2019] during any oxygen therapy, the inspired O2 concentration is usually adapted to a pre-set SpO2 target-range of 92-96% in patients without hypercapnia risk, and of 88-92% if a risk of hypercapnia is present [O'Driscoll et al, 2017; Beasley et al, 2015]. In most institutions, the standard of care is to manually adapt the FiO2, although patients frequently have a SpO2 value outside the target range.

A new closed loop oxygen controller designed for HFNO was recently developed (Hamilton Medical, Bonaduz, Switzerland). The clinician sets SpO2 targets, and the software option adjusts FiO2 to keep SpO2 within the target ranges. The software option offers some alarms on low and high SpO2 and high FiO2. Given the capability, on the one hand, to quickly increase FiO2 in patients developing sudden and profound hypoxia, and, on the other hand, of automatically preventing hyperoxia in patients improving their oxygenation, such a system could be particularly useful in patients treated with HFNO.

A short-term (4 hours vs 4 hours) crossover study indicated that this technique improves the time spent within SpO2 pre-defined target for ICU patients receiving high-flow nasal oxygen therapy [Roca et al, 2022]. Due to its simplicity, HFNO is increasingly used outside the ICU during transport and in the Emergency Room (ER). This environment poses specific challenges, as patients may deteriorate very quickly and depending on patient's flow, healthcare providers can easily be overwhelmed. We thus propose to evaluate closed loop controlled HFNO in ER patients.

The hypothesis of the study is that closed loop oxygen control increases the time spent within clinically targeted SpO2 ranges and decreases the time spent outside clinical target SpO2 ranges as compared to manual oxygen control in ER patients treated with HFNO.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the ER
* Requiring NHFO
* Requiring FiO2 ≥ 30% to keep SpO2 in the target ranges defined by the clinician
* Aged over 18 years
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation
* In case that the consent is given by the relative, patient consent will be requested as soon as the patient will be able to provide informed written consent

Exclusion Criteria:

Patients who fulfil any of the following exclusion criteria are not eligible for study participation:

* Patient with indication for immediate CPAP, NIV, or invasive mechanical ventilation
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h
* Low quality on the SpO2 measurement using finger and ear sensor (quality index below 60% on the Massimo SpO2 sensor, which is displayed by a red or orange color bar)
* Severe acidosis (pH ≤ 7.30)
* Pregnant woman
* Patients deemed at high risk for need of mechanical ventilation within the next 12 hours
* Chronic or acute dyshemoglobinemia: methemoglobin, CO poisoning, sickle cell disease
* Tracheotomized patient
* Formalized ethical decision to withhold or withdraw life support
* Patient under guardianship
* Patient deprived of liberties
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of acute respiratory failure

Post enrollment exclusion criteria

* Apparition of a persistent low quality SpO2 signal
* Need for an emergent intubation
* Discharge from ER

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in optimal SpO2 range | 6 hours
  The optimal SpO2 range will be defined according to the SpO2 targets determined by the clinician.

SECONDARY OUTCOMES:
Percentage of time with SpO2 signal available | 6 hours
  Time with SpO2 signal available
Percentage of time with SpO2 below target range | 6 hours
  SpO2 values below the optimal range
Percentage of time with SpO2 above target range | 6 hours
  SpO2 values above the optimal range
Percentage of time with SpO2 outside optimal range | 6 hours
  SpO2 values outside the optimal range
Percentage of time with with FiO2 below 40% | 6 hours
  Duration of time with FiO2 < 40 %
Percentage of time with with FiO2 above 60% | 6 hours
  Duration of time with FiO2 > 60 %
Percentage of time with with FiO2 = 100% | 6 hours
  Duration of time with FiO2 = 60 %
Mean SpO2/FiO2 | 6 hours
  Mean SpO2/FiO2
Number of events with SpO2 below of target range (duration >10 s) | 6 hours
  Frequency of events with SpO2 below of target range (duration >10 s)
Number of events with SpO2 below of target range (duration >60 s) | 6 hours
  Frequency of events with SpO2 below of target range (duration >60 s)
Number of events with SpO2 below the predefined low SpO2 emergency limit | 6 hours
  Frequency of events with SpO2 below of the predefined low SpO2 emergency limit
Number of events with SpO2 above the predefined low SpO2 emergency limit | 6 hours
  Frequency of events with SpO2 above of the predefined low SpO2 emergency limit
Total oxygen use | 6 hours
  Amount of additional oxygen use

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Guven, Associate prof, Principal Investigator — Basaksehir Cam Sakura city Hospital, Istanbul
Locations (2):
- Turkey (Türkiye) (2):
  - Başakşehir Çam & Sakura City Hospital, Istanbul
  - Dr.Suat Seren Chest Diseasees Hospital, Izmir

REFERENCES:
- [Background] Sandal O, Ceylan G, Topal S, Hepduman P, Colak M, Novotni D, Soydan E, Karaarslan U, Atakul G, Schultz MJ, Agin H. Closed-loop oxygen control improves oxygenation in pediatric patients under high-flow nasal oxygen-A randomized crossover study. Front Med (Lausanne). 2022 Nov 16;9:1046902. doi: 10.3389/fmed.2022.1046902. eCollection 2022. PMID 36465920
- [Background] Roca O, Caritg O, Santafe M, Ramos FJ, Pacheco A, Garcia-de-Acilu M, Ferrer R, Schultz MJ, Ricard JD. Closed-loop oxygen control improves oxygen therapy in acute hypoxemic respiratory failure patients under high flow nasal oxygen: a randomized cross-over study (the HILOOP study). Crit Care. 2022 Apr 14;26(1):108. doi: 10.1186/s13054-022-03970-w. PMID 35422002
- [Background] Dijkman KP, Goos TG, Dieleman JP, Mohns T, van Pul C, Andriessen P, Kroon AA, Reiss IK, Niemarkt HJ. Predictive Intelligent Control of Oxygenation in Preterm Infants: A Two-Center Feasibility Study. Neonatology. 2023;120(2):235-241. doi: 10.1159/000527539. Epub 2022 Dec 8. PMID 36481622
- [Background] O'Driscoll BR, Kirton L, Weatherall M, Bakerly ND, Turkington P, Cook J, Beasley R. Effect of a lower target oxygen saturation range on the risk of hypoxaemia and elevated NEWS2 scores at a university hospital: a retrospective study. BMJ Open Respir Res. 2024 Feb 29;11(1):e002019. doi: 10.1136/bmjresp-2023-002019. PMID 38423953